CLINICAL TRIAL: NCT02314455
Title: Esophageal Absorption in Eosinophilic Esophagitis
Brief Title: Esophageal Absorption in EoE
Acronym: EoE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early analysis showed negative results. It was decided to halt the study.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David A. Katzka, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-009092
Record Dates: First submitted 2014-11-10; First posted 2014-12-11 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; EoE; dysphagia
MeSH Terms: conditions — Eosinophilic Esophagitis; Deglutition Disorders | interventions — Xylose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- D-xylose, water, honey (Experimental): * 25 grams of D-xylose
  * 10 cc of water
  * 2 teaspoons of honey
  Interventions: Other: D-xylose

INTERVENTIONS:
Other: D-xylose — There will be four patient groups analyzed. Ten patients each, 10 with active eosinophilic esophagitis defined by consensus guidelines, 20 patients in histologic remission (10 by steroids and 10 by diet) and 10 control volunteers will be studied. Patients who have consented to the trial will be scheduled at the Clinical Research Unit (CRU) Patients will report to Charlton 7 the CRU, having their height, weight, blood pressure and temperature recorded. Subjects can choose to either have a saline lock IV placed or have their bloods drawn 3 separate times. They will receive 25 grams of D-xylose orally. The D-xylose will be mixed in 10 cc of water with 2 teaspoons of honey. D-xylose serum levels will be drawn at 5 and 10 and 60 minutes.
  Other Names: Eosinophilic esophagitis; Absorption study

SUMMARY:
To determine how the esophagus in active and inactive stages of eosinophilic esophagitis tranmit fluids.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 80 with eosinophilic esophagitis diagnosed by a combination of compatible symptoms, endoscopic findings, histology, and lack of response to proton pump inhibitors or negative pH study
* endoscopy with esophageal and duodenal biopsies within two weeks of performance of this study
* Patients between the ages of 18 and 80 with eosinophilic esophagitis diagnosed by a combination of compatible symptoms, endoscopic findings, histology, and lack of response to proton pump inhibitors or negative pH study, and are now in histologic remission( <15phf) by the use of steroids or the six food elimination diet.
* Volunteers will be selected for not having any history of esophageal symptoms

Exclusion Criteria:

* Vulnerable populations, such as those with diminished mental acuity, will be excluded.
* Patients taking Nsaids within 48 hours of the d-xylose testing
* artificial sweeteners within 48 hours of the d-xylose testing
* History of IBD
* Currently smoking or history of smoking
* History of Celiac disease
* Bacterial overgrowth,
* motility disorders
* other diffuse small bowel diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Reliability of the d-xylose testing defined by the serum levels | 1 year
  D-xylose serum levels will be drawn at 5 and 10 and 60 minutes. D-xylose levels will be compared between the patients with active EOE and healthy controls using the Wilcoxon rank sum test.

SECONDARY OUTCOMES:
D-xylose testing compared to endoscopy/biopsy findings. | 1 year
  Histologic parameters will include grading of spongiosis as an indicator of dilated intercellular spaces which will be correlated to serum levels of D-xylose.

CONTACTS AND LOCATIONS:
Overall Officials: David Katzka, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States